CLINICAL TRIAL: NCT05828381
Title: A Prospective, Single-arm Multicenter Clinical Trial of Envafolimab Combined With Abraxane and Cisplatinas in Resectable Esophageal Squamous Cell Cancer
Brief Title: Envafolimab Combined With Abraxane and Cisplatinas as Neoadjuvant Treatment for Resectable Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mingqiang Kang
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Immunotherapy;Envafolimab; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — envafolimab; Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab combination with Abraxane and cisplatin (Experimental): Arm description：Envafolimab:300mg,sc,d1,q3w; for a total of 2 cycles. Chemotherapy： Abraxane + Cisplatin Abraxane :100mg/m2,ivgtt, D1、D8,q3w ,for a total of 2 cycles. Cisplatin : 75 mg/m 2 vigtt D1 , q3w , for a total of 2 cycles.
  Interventions: Drug: Envafolimab; Drug: Abraxane; Drug: Cisplatin

INTERVENTIONS:
Drug: Envafolimab — 300mg,sc,d1,q3w; for a total of 2 cycles.
Drug: Abraxane — 100mg/m2,ivgtt, D1、D8,q3w ,for a total of 2 cycles
Drug: Cisplatin — 75 mg/m2 vigtt D1 , q3w , for a total of 2 cycles

SUMMARY:
Big breakthroughs have been made in the combination therapy of immune checkpoint inhibitors when it comes to the neoadjuvant therapy of esophageal cancer. Several studies, such as Cross, have shown that although preoperative adjuvant chemoradiotherapy could improve the local control rate of lesions, the incidence of distant metastasis still remains high in the long term. Compared with preoperative adjuvant chemoradiotherapy, the treatment of combination with immunotherapy has shown a lot of advantages such as shorter hospital stay, fewer complications and lower cost, which may replace preoperative chemotherapy or chemoradiotherapy for esophageal cancer as a new treatment .This is a single-arm, exploratory phase II clinical study to evaluate the efficacy and safety of Envafolimab combination with Abraxane and cisplatin as preoperative neoadjuvant therapy for patients with resectable esophageal squamous cell carcer. In the study, all subjects meeting enrollment criteria will receive 2 cycles of neoadjuvant therapy with Envafolimab combined with Abraxane and cisplatin as scheduled. Around 4-6 weeks after the last neoadjuvant therapy, they will receive radical surgery. Evaluation will be conducted after the completion of the surgical cycle to determine the pathological complete response rate , R0 resection rate and major pathological response rate of these treated patients.

The objective is To evaluate the efficacy and safety of Enbrelizumab in combination with Abraxane and cisplatin for preoperative neoadjuvant therapy in patients with resectable esophageal squamous cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily joins this study and is able to sign the informed consent form with good compliance;
* 18-75 years of age (at the time of signing the informed consent);
* ECOG score 0-1;
* Expected survival ≥ 12 weeks;
* Patients with confirmed diagnosis of esophageal squamous cell carcinoma by histopathologic examination of primary tumor biopsy, who are definitely diagnosed with clinical stage of esophageal cancer by CT or MRI or color Doppler ultrasound or PET-CT or endoscopic ultrasonography T1-3N1-3M0 or T3N0M0 (AJCC 8 th) and are suitable for treatment with this study protocol as assessed by the investigator.
* No previous anti-tumor therapy, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc . However, exploratory thoracotomy, mediastinoscopy, excisional biopsy, or similar surgical procedures performed to confirm the diagnosis, staging, and surgical treatment of esophageal cancer are acceptable.
* Adequate major organ function meeting the following criteria:1) Hematology (without blood transfusion or hematopoietic stimulating factor drugs within 14 days): hemoglobin (Hb) ≥ 90 g/L; absolute neutrophil count (ANC) ≥ 1.5 × 10 9/L; platelet (PLT) ≥ 100 × 10 9/L;Biochemistry: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; serum total bilirubin (TBIL) ≤ 1.5 × ULN (in subjects with Gilbert 's syndrome, ≤ 3 × ULN); serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min;3)Urine routine: urine protein < 2 +; if urine protein ≥ 2 +, 24-hour urine protein quantification must show protein ≤ 1 g;4) Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;5) Euthyroid defined as thyroid stimulating hormone (TSH) within normal limits. If baseline TSH is out of normal range, subjects with total T3 (or FT3) and FT4 within normal range can also be enrolled;
* Adequate organ function as judged clinically by the physician ;
* Subjects of childbearing potential must use adequate contraception during this study and for 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating.

Exclusion Criteria:

* Suffered from other malignant tumors within 5 years before the start of treatment in this study;
* Patients with tumor invasion of cervical esophagus or upper thoracic segment requiring laryngectomy;
* Patients with high risk of bleeding or perforation due to tumor obvious invasion of the organs adjacent to the esophageal lesion (major artery or trachea) or patients with fistula;
* Subjects with any severe or uncontrolled medical conditions;
* Poor blood pressure control (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg);
* Patients with poorly controlled cardiac clinical symptoms or diseases such as: (1) NYHA2 or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* The subject had an active infection or unexplained fever during screening and prior to initial administration (if the subject had fever due to the tumor, as determined by the investigator, he could be enrolled);
* Previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc.;
* Patients with acute or chronic active Hepatitis B ;
* A history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
* Poor diabetes control;
* Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
* Study participants who received major surgical treatment, open biopsy, or significant traumatic injury within 28 days before the start of treatment or a wound or fracture that has not healed for a long time;
* Severe arteriovenous thrombosis events;
* Those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders;
* Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage;
* Subjects with known central nervous system metastatic and/or cancerous meningitis;
* Study the history of live attenuated vaccine vaccination within 14 days prior to the start of treatment or planned live attenuated vaccine vaccination during the study period;
* Active autoimmune diseases requiring systemic treatment have occurred within 2 years prior to the initiation of the study treatment, other than alternative therapies;
* Diagnosed with immunodeficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy;
* People with a history of active tuberculosis;
* Participating in or having participated in other clinical investigators within 4 weeks prior to study initiation;
* Previous treatment with other PD-1/PD-L1 inhibitors could not be included in the group; the subject known to have a prior allergy to macromolecular protein preparations;
* Those who are known to be allergic to the active ingredients or excipients of the drug in this study, such as Envollizumab, albumin paclitaxel and cisplatin;
* Subjects who, in the investigator's judgment, have a concomitant medical condition that seriously endangers subjects' safety or interferes with the completion of the study, or who are deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The pathological complete response rate | 1 year

SECONDARY OUTCOMES:
The R0 resection rate | 1 year
The major pathological response rate | 1 year
The disease free survival rate | 1 year

IPD SHARING:
Plan to Share IPD: No